CLINICAL TRIAL: NCT00454337
Title: Randomized Non-inferiority Study Comparing a Strategy Maintaining Current Enfuvirtide-based Antiretroviral Therapy to a Strategy Replacing Enfuvirtide by an Integrase Inhibitor (Raltegravir) in HIV-1 Infected Subjects With Plasma Hiv-1 RNA Levels Below 400 Copies Per ml.ANRS 138 EASIER
Brief Title: Efficacy and Tolerance of the Switch From Enfuvirtine to Raltegravir in Antiretroviral Therapy Regimen in HIV Patients With Undetectable Viral Load
Acronym: EASIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-000162-20; ANRS 138 EASIER
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; enfuvirtide; raltegravir; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensification arm (Experimental): emtricitabine/TDF + efavirenz or lopinavir/ritonavir + enfuvirtide
  Interventions: Drug: FTC/TDF + EFV or LPV/R +T20
- Standard arm (Active Comparator): emtricitabine/TDF + efavirenz or lopinavir/ritonavir
  Interventions: Drug: FTC/TDF + EFV or LPV/R

INTERVENTIONS:
Drug: FTC/TDF + EFV or LPV/R +T20 — emtricitabine 200mg/TDF 300mg (1 pill per day) + efavirenz 600mg (1 pill per day) or lopinavir/ritonavir (3 pills twice a day) + enfuvirtide 90mg twice a day
  Arms: Intensification arm
Drug: FTC/TDF + EFV or LPV/R — emtricitabine 200mg/TDF 300mg (1 pill per day) + efavirenz 600mg (1 pill per day) or lopinavir/ritonavir (3 pills twice a day)
  Arms: Standard arm

SUMMARY:
Switching from enfuvirtide to raltegravir in the treatment of HIV-infected patients who sustain viral suppression with a combination therapy including enfuvirtide (or : with an enfuvirtide-based combination therapy)

DETAILED DESCRIPTION:
In patients who have failed under the three main classes of antiretroviral agents (NRTI, NNRTI and PI) and in whom the control of viral replication in the plasma has ultimately been achieved with enfuvirtide, the aim is to sustain this virological success for as long as possible to thus enable satisfactory immune reconstitution, avoid further accumulation of viral mutations conferring resistance to the drugs and protect the patient from the risk of opportunistic disease and death.

Indeed, enfuvirtide is the lead compound in the new class of antiretroviral drugs which inhibit the fusion of HIV-1 virus with its target cell. Its in vivo efficacy was demonstrated during the pivotal studies TORO 1 and 2. Despite its efficacy, maintaining long-term treatment with enfuvirtide is nonetheless difficult for patients because of the constraints related to twice-daily subcutaneous parenteral injections. Furthermore, these subcutaneous injections are associated with inflammatory reactions at the injection site in 98 per cent of patients, without any reduction in frequency or severity over time. It is thus critical for patients who are well controlled by enfuvirtide to be able to simplify their treatment by replacing enfuvirtide with another active compound taken by mouth, which would enable maintenance of the virological response and acceptable safety in patients who have usually failed under the three main classes of antiretroviral drugs. A new antiviral compound, viral integrase inhibitor called raltegravir, could be proposed instead of enfuvirtide.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV-1 infection
* Treatment with a well-tolerated combination of antiretroviral drugs unchanged for at least 3 months, including enfuvirtide
* Absence of any uncontrolled opportunistic disease
* No restrictions on CD4 lymphocyte levels
* Plasma HIV-1 RNA below 400 copies per ml for at least 3 months (at least two consecutive tests below 400 copies per ml prior to inclusion in the study, not including that on W -4)
* For women of childbearing age, use of mechanical contraception during any sexual intercourse and negative pregnancy test (plasma ß HCG) at W -4

Exclusion Criteria:

* HIV-2 infection
* Plasma HIV-1 RNA levels above 400 copies/ml on one occasion during the 3 months prior to screening (or the pre-inclusion visit at W -4)
* Poor compliance with antiretroviral therapy current at W -4
* Current treatment with an investigational drug (except cohort ATU)
* Patient previously treated with an integrase inhibitor in the context of a clinical study
* Woman who is pregnant or likely to become so, is breastfeeding or refuses to use contraception
* Multiple drug therapy ongoing or necessary in the foreseeable future for Kaposi's disease or lymphoma
* Treatment with interferon ongoing or necessary in the foreseeable future for chronic hepatitis B or C
* Acute hepatitis whatever the case, or decompensated cirrhosis
* Current treatment with interferon, interleukin or anti-HIV vaccine
* Any condition (including, but not limited to, the consumption of alcohol or drugs) which might, in the investigator's opinion, compromise the safety of treatment and/or patient compliance with the protocol
* Significant biological abnormalities (hemoglobin below 8g per dl, polynuclear neutrophils below 750 per mm3, platelets below 50,000 per mm3, serum creatinine above 3 times the level deemed normal by the laboratory (N), ASAT or ALAT above 5N, serum lipase above 2N) and total bilirubin above 2N (except if the patient is receiving atazanavir or indinavir)
* Concomitant treatments including one or more compounds interacting with UGT1A1

  * anti-infective agents: rifampicin/rifampin
  * psychotropic/anti-epileptic drugs: phenytoin, phenobarbital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
comparison of the proportions of virologic failure, defined as two consecutive pVL above 400 cp per ml, through 24 weeks in enfuvirtide-maintained arm versus raltegravir arm | W24

SECONDARY OUTCOMES:
comparison of time to onset of virologic failure | W24 and W48
proportions of pts with pVL under 50 and 400 cp per ml respectively at week 24 and week 48 ; | W24 & W48
plasma viral mutations in the event of virologic failure, compared to HIV-DNA archived mutations at baseline; | virologic failure
change in CD4 levels | between W0 and W48
incidence of HIV-related events | between W0 and W48
drug plasma and male genital tract pharmacokinetics; | W24 & W48
incidence and type of adverse events, including adverse reactions | between W0 & W48
proportions of discontinuing allocated treatment strategy | between W0 & W48
quality of life and adherence | W4, W12, W24 and W48
morphological and metabolic disorders outcome | between W0 & W48

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie De Castro, MD, Principal Investigator — AP-HP Hopital Saint Louis Paris; Jean M Molina, MD, Principal Investigator — AP-HP Hopital saint Louis Paris; Jean P Aboulker, MD, Study Chair — INSERM SC10 Villejuif France
Locations (1):
- Service des maladies infectieuses et tropicales Hopital Saint Louis, Paris, France

REFERENCES:
- [Result] Goldwirt L, Braun J, de Castro N, Charreau I, Barrail-Tran A, Delaugerre C, Raffi F, Lascoux-Combe C, Aboulker JP, Taburet AM, Molina JM. Switch from enfuvirtide to raltegravir lowers plasma concentrations of darunavir and tipranavir: a pharmacokinetic substudy of the EASIER-ANRS 138 trial. Antimicrob Agents Chemother. 2011 Jul;55(7):3613-5. doi: 10.1128/AAC.01827-10. Epub 2011 May 16. PMID 21576452
- [Result] Barau C, Delaugerre C, Braun J, de Castro N, Furlan V, Charreau I, Gerard L, Lascoux-Combe C, Molina JM, Taburet AM. High concentration of raltegravir in semen of HIV-infected men: results from a substudy of the EASIER-ANRS 138 trial. Antimicrob Agents Chemother. 2010 Feb;54(2):937-9. doi: 10.1128/AAC.01261-09. Epub 2009 Dec 7. PMID 19995925
- [Result] Delaugerre C, Charreau I, Braun J, Nere ML, de Castro N, Yeni P, Ghosn J, Aboulker JP, Molina JM, Simon F; ANRS 138 study group. Time course of total HIV-1 DNA and 2-long-terminal repeat circles in patients with controlled plasma viremia switching to a raltegravir-containing regimen. AIDS. 2010 Sep 24;24(15):2391-5. doi: 10.1097/QAD.0b013e32833d214c. PMID 20683319
- [Result] Boulet T, Pavie J, Charreau I, Braun J, Reynes J, Morlat P, Piroth L, Spire B, Molina JM, Aboulker JP; Easier-Anrs 138 Study Group. Impact on health-related quality of life of a switch from enfuvirtide to raltegravir among multidrug-resistant HIV-1-infected patients: a randomized open-label trial (EASIER-ANRS 138). HIV Clin Trials. 2010 Sep-Oct;11(5):283-93. doi: 10.1310/hct1105-283. PMID 21126958
- [Result] Gallien S, Delaugerre C, Charreau I, Braun J, Boulet T, Barrail-Tran A, de Castro N, Molina JM, Kuritzkes DR. Emerging integrase inhibitor resistance mutations in raltegravir-treated HIV-1-infected patients with low-level viremia. AIDS. 2011 Mar 13;25(5):665-9. doi: 10.1097/QAD.0b013e3283445834. PMID 21326075
- [Result] Gallien S, Braun J, Delaugerre C, Charreau I, Reynes J, Jeanblanc F, Verdon R, de Truchis P, May T, Madelaine-Chambrin I, Aboulker JP, Molina JM; EASIER ANRS 138 Study Group. Efficacy and safety of raltegravir in treatment-experienced HIV-1-infected patients switching from enfuvirtide-based regimens: 48 week results of the randomized EASIER ANRS 138 trial. J Antimicrob Chemother. 2011 Sep;66(9):2099-106. doi: 10.1093/jac/dkr269. Epub 2011 Jun 28. PMID 21712241
- [Result] Delaugerre C, Braun J, Charreau I, Delarue S, Nere ML, de Castro N, May T, Marchou B, Simon F, Molina JM, Aboulker JP; ANRS 138-EASIER study group. Comparison of resistance mutation patterns in historical plasma HIV RNA genotypes with those in current proviral HIV DNA genotypes among extensively treated patients with suppressed replication. HIV Med. 2012 Oct;13(9):517-25. doi: 10.1111/j.1468-1293.2012.01002.x. Epub 2012 Mar 14. PMID 22416781
- [Derived] de Castro N, Braun J, Charreau I, Lafeuillade A, Viard JP, Allavena C, Aboulker JP, Molina JM; EASIER ANRS 138 study group. Incidence and risk factors for liver enzymes elevations in highly treatment-experienced patients switching from enfuvirtide to raltegravir: a sub-study of the ANRS-138 EASIER trial. AIDS Res Ther. 2016 Apr 2;13:17. doi: 10.1186/s12981-016-0101-3. eCollection 2016. PMID 27042193
- [Derived] De Castro N, Braun J, Charreau I, Pialoux G, Cotte L, Katlama C, Raffi F, Weiss L, Meynard JL, Yazdanpanah Y, Delaugerre C, Madelaine-Chambrin I, Aboulker JP, Molina JM; EASIER ANRS 138 study group. Switch from enfuvirtide to raltegravir in virologically suppressed multidrug-resistant HIV-1-infected patients: a randomized open-label trial. Clin Infect Dis. 2009 Oct 15;49(8):1259-67. doi: 10.1086/605674. PMID 19757993